CLINICAL TRIAL: NCT03786705
Title: The Relationship of Delta Shock Index With the Requirement of Blood Transfusion and Clinical Outcome of Adult Trauma Patients
Brief Title: Delta Shock Index in Predicting Massive Transfusion
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG8G1301
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Trauma Patients Received Blood Transfusion ≥ 10 U; Trauma Patients Had Not Received Blood Transfusion ≥ 10 U

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma patients' SBP ≥ 90 mm Hg with EMS: Only patients who were transferred by emergency medical service from the accident site with a systolic blood pressure ≥ 90 mm Hg at the ER were included in this study. The enrolled trauma patients divided into 2 groups, those who had received blood transfusion ≥ 10 U (massive transfusion) and those who had not (non-massive transfusion).
  Interventions: Other: Massive transfusion; Other: Non-Massive Transfusion

INTERVENTIONS:
Other: Massive transfusion — Trauma patients who had received blood transfusion≥10 U
Other: Non-Massive Transfusion — Trauma patients who had received blood transfusion<10 U

SUMMARY:
Background: To determine the performance of delta shock index (ΔSI), a change in shock index (SI) upon arrival at the emergency room (ER) from that in the field in predicting the need for massive transfusion (MT) among adult trauma patients with stable blood pressure.

Methods: This study included data from all trauma patients aged 20 years and above who were hospitalized from January 1, 2009 to December 31, 2016 and was obtained from the registered trauma database of the hospital. Only patients who were transferred by emergency medical service from the accident site with a systolic blood pressure ≥ 90 mm Hg at the ER were included in this study. The 7,957 enrolled trauma patients were divided into 2 groups, those who had received blood transfusion ≥ 10 U (MT, n = 82) and those who had not (non-MT, n = 7,875). The odds ratios with 95% confidence intervals for associated patient conditions and the odds of need for MT by a given ΔSI were measured. The plot of specific receiver operating characteristic (ROC) curves was used to evaluate the best cutoff point that could predict the patient's probability of receiving MT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were transferred by emergency medical service (EMS) from the field of accident and had a stable blood pressure (SBP ≥ 90 mmHg) at the ER were included

Exclusion Criteria:

* Patients who were transferred from other hospitals or arrived by private vehicles.
* Patients who had incomplete data
* Patients who had an unstable blood pressure (SBP < 90 mmHg) upon arrival at the ER were also excluded

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hospitalized trauma patients aged 20 years and above from January 1, 2009 to December 31, 2016 from the registered trauma database of the hospital.
Sampling Method: Probability Sample
Enrollment: 7957 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
in-hospital mortality | up to 5 months
  To measure the outcome of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan